CLINICAL TRIAL: NCT04698122
Title: Costituzione Della Biobanca Del Microbiota Intestinale e Salivare Umano: Dalla Disbiosi Alla Simbiosi
Brief Title: Establishment of the Human Intestinal and Salivary Microbiota Biobank- Diabetes
Acronym: BIOMIS-Diab
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Institute of Biomembranes, Bioenergetics and Molecular Biotechnologies (Other); University Of Perugia (Other); University of Bari Aldo Moro (Other); University of Salento (Other); Istituti Tumori Giovanni Paolo II (Network)
Responsible Party: Sponsor
Other Study IDs: BIOMIS-Diab
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Microbioma biobank; Biological human samples; diabetes; Meta-omics approaches; Microbiota-pathology relationship
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Surveys and Questionnaires; Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — faeces, saliva, blood, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- type 1 diabetes: Patients with type 1 diabetes
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- type 2 diabetes: Patients with type 2 diabetes
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- Healthy volunteers: Healthy volunteers
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination

INTERVENTIONS:
Other: Biological sample collection — Collection of faeces, urine, saliva, and blood for biobanking, to evaluate the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile, and to perform routine screening
Other: Questionnaire — Anamnestic questionnaire, 3-day food questionnaire, Food Frequency Questionnaire
Other: Medical examination — Blood pressure measurement, abdominal and thoracic physical examination

SUMMARY:
This is a prospective, clinical, monocentric study aimed to collect biological samples and study microbiota from subjects suffering from type 1 diabetes mellitus, subjects suffering from type 2 diabetes mellitus and from healthy volunteers. Microbiota is a complex consortium of microorganisms, located at the mucosal level (in particular intestinal, oral and vaginal) having a key role in human health and in the onset of several diseases. Microbiota alterations have been found in several diseases (gastrointestinal, metabolic, renal, oncological, gynaecological).

The study will allow to:

* Provide biological samples (faeces, saliva, blood, urine) from healthy volunteers and patients suffering with diabetes mellitus 1 and 2 to the first Italian microbiota biobank;
* Study microorganisms using different in vitro and in vivo techniques;
* Study the link between the microbiota and the disease. This study is part of the BIOMIS project (Project Code: ARS01_01220), presented as part of the "Avviso per la presentazione di progetti di ricerca industriale e sviluppo sperimentale nelle 12 aree di specializzazione individuate dal PNR 2015-2020" and admitted to funding under the National Operational Program "Ricerca e Innovazione" 2014-2020 by directorial decree of MIUR - Department for Higher Education and Research - n. 2298 of 12 September 2018. BIOMIS includes several clinical studies that enrol patients with different pathologies to collect and store biological samples and study microbiota.

DETAILED DESCRIPTION:
The primary aim of this monocentric study is to populate the first national microbioma biobank with biological samples (fecal, salivary, urinary and blood samples) subjects suffering from diabetes mellitus 1 and 2, and healthy volunteers.

The secondary aim is the characterization of microorganisms of the biobank and study of the microbiota-pathology relationship using meta-omics, in vitro and in vivo approaches, The study plans to enrol 75 subjects at University of Perugia, according to the inclusion/exclusion criteria. The study participation is voluntary, and the subjects have the right to withdraw from the study at any time and for any reason.

During the study, 3 visits are planned:

* Visit 0 (V0), including description of the objectives and procedures study, signature written informed consent, inclusion/exclusion criteria evaluation, medical examination (blood pressure measurement, abdominal and thoracic physical examination), filling in of the anamnestic questionnaire, delivery of kits for the collection of fecal, salivary and urinary material to be reported at Visit 1 and delivery of a 3-day food diary, to be completed autonomously in the days preceding the Visit 1.
* Visit 1 (V1) - at least 4 days after V0, including delivery of the of the collected biological material (feces, saliva, urine), and of a 3-day food diary, filling in of the new signs and symptoms anamnestic questionnaire and blood sampling by medical staff.
* Telephone evaluation: administration of a "Food Frequency Questionnaire" to assess the subjects' alimentary habits.

Standard Operative Procedures (SOP) for samples storing, transport and processing will be adopted to ensure samples stability and grant results validity and quality.

Following collections, samples will be processed in different aliquots that will be used for:

* routine screening;
* storage in the first Italian human microbiote biobank (I.R.C.C.S. - Istituto Tumori "Giovanni Paolo II", Bari);
* evaluation of the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile.

Furthermore, molecular characterization of pathogenic microorganisms and pathogenic biotypes (pathovars) of commensal species of subjects with selected pathologies will be conducted.

Part of the biological material will be used for animal studies on the physiopathological role of the human intestinal microbiota transplanted into mouse models of pathology and Germ-free mouse models (specific animal study protocol developed).

The study foresees no more than minimal risk associated with blood sampling procedures. All the necessary measures to avoid any risks / inconveniences resulting from participation of the subject under study will be taken.

The study is compliant with Good Clinical Practice. Study protocol and all related documents have been approved by approved by the Independent Ethics Committees (IEC) of the involved clinical sites.

To ensure the protection and confidentiality of the participants' data, all study activities will be carried out in accordance with the European General Data Protection Regulation, Regulation (EU) 2016/679, which repeals Directive 95/46/EC.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEERS

* healthy subjects aged between 18 and 60 years
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

TYPE 1/TYPE 2 DIABETES

* subjects with type 1 diabetes aged between 18 and 50 years, type 2 diabetes aged between 18 and 65 years
* creatinine clearance > 60 mL / min
* Normoalbuminurics (ACR <30 mg / g)
* Absence of diabetic retinopathy
* DM duration <5 years
* Not being treated with metformin
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

Exclusion Criteria:

HEALTHY VOLUNTEERS

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Healthcare workers
* Operators work with animals
* Psychiatric conditions that reduce protocol compliance.

TYPE 1/TYPE 2 DIABETES

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent emergence of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke) occurred in the last 3 years
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Psychiatric conditions that reduce protocol compliance.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 and 2 diabetes attending the clinical centres involved in the study.
  Healthy volunteers will be recruited by invitation. Enrolled subjects must not have any family relationship and hierarchical subordination with the hospitals in which biological samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Biological samples collection for establishment of the first National Microbiome Biobank | through study completion, an average of 1 year
  Recruitment of 75 subjects (type 1 diabetes, type 2 diabetes patients and healthy volunteers) to collect biological samples for establishment of the first National Microbiome Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Reboldi, MD, Principal Investigator — University Of Perugia
Locations (1):
- Università degli Studi di Perugia - Dipartimento di Medicina, S.C. Endocrinologia e Malattie del Metabolismo-Azienda Ospedaliera di Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu F, Han W, Zhan G, Li S, Jiang X, Wang L, Xiang S, Zhu B, Yang L, Luo A, Hua F, Yang C. Abnormal gut microbiota composition contributes to the development of type 2 diabetes mellitus in db/db mice. Aging (Albany NY). 2019 Nov 23;11(22):10454-10467. doi: 10.18632/aging.102469. Epub 2019 Nov 23. PMID 31760385
- [Background] Bordalo Tonucci L, Dos Santos KM, De Luces Fortes Ferreira CL, Ribeiro SM, De Oliveira LL, Martino HS. Gut microbiota and probiotics: Focus on diabetes mellitus. Crit Rev Food Sci Nutr. 2017 Jul 24;57(11):2296-2309. doi: 10.1080/10408398.2014.934438. PMID 26499995
- [Background] Munoz-Garach A, Diaz-Perdigones C, Tinahones FJ. Gut microbiota and type 2 diabetes mellitus. Endocrinol Nutr. 2016 Dec;63(10):560-568. doi: 10.1016/j.endonu.2016.07.008. Epub 2016 Sep 12. English, Spanish. PMID 27633134
- [Background] Tilg H, Moschen AR. Microbiota and diabetes: an evolving relationship. Gut. 2014 Sep;63(9):1513-21. doi: 10.1136/gutjnl-2014-306928. Epub 2014 May 15. PMID 24833634